CLINICAL TRIAL: NCT03017404
Title: A Dose Increase Finding Study of Doxorubicin Hydrochloride Liposome Injection in Neoadjuvant Chemotherapy for Patients With Locally Advanced Breast Cancer
Brief Title: A Dose Increase Finding Study of Doxorubicin Hydrochloride Liposome Injection for Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-BC-02
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- treatment group:35 mg/m(2) (Experimental): Doxorubicin Hydrochloride Liposome injection combination with cyclophosphamide and sequential treatment of docetaxel, 4 cycles (each cycle is 21 days) of chemotherapy
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Cyclophosphamide; Drug: docetaxel
- treatment group:40 mg/m(2) (Experimental): Doxorubicin Hydrochloride Liposome injection combination with cyclophosphamide and sequential treatment of docetaxel, 4 cycles (each cycle is 21 days) of chemotherapy
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Cyclophosphamide; Drug: docetaxel
- treatment group:45 mg/m(2) (Experimental): Doxorubicin Hydrochloride Liposome injection combination with cyclophosphamide and sequential treatment of docetaxel, 4 cycles (each cycle is 21 days) of chemotherapy
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Cyclophosphamide; Drug: docetaxel
- treatment group:50 mg/m(2) (Experimental): Doxorubicin Hydrochloride Liposome injection combination with cyclophosphamide and sequential treatment of docetaxel, 4 cycles (each cycle is 21 days) of chemotherapy
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection; Drug: Cyclophosphamide; Drug: docetaxel

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome Injection
Drug: Cyclophosphamide
Drug: docetaxel

SUMMARY:
To study the maximum tolerated dose of Doxorubicin Hydrochloride Liposome Injection combination with cyclophosphamide and sequential treatment of docetaxel for patients with locally advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Female patients newly diagnosed breast cancer≥18 and ≤70 years of age;
* Karnofsky performance status≥70 and measurable or evaluable;
* Stages Ⅲa-ⅢC;
* Baseline left ventricular ejection fraction (LVEF) ≥ 50%;
* Adequate marrow function (WBC count> 4.0×10(9)/L, neutrophil> 2.0×10(9)/L, platelet count > 100×10(9)/L，hemoglobin > 90g/L );
* AST and ALT ≤1.5× institutional upper limit of normal, alkaline phosphatase
* ≤2.5×institutional upper limit of normal，bilirubin ≤institutional upper limit of normal;
* Serum creatinine ≥ 44µmol/L and ≤ 133 µmol/L;
* Expected lifetime ≥ 12 months;
* Pregnancy tests of reproductive age women is negative;
* All patients provided written informed consent.

Exclusion Criteria:

* Distant metastasis;
* Severe heart failure (NYHA grade II or higher);
* Active and uncontrolled severe infection;
* Hypersensitivity to anthracycline therapy or a history of severe hypersensitivity reactions to products containing liposomal doxorubicin and docetaxel;
* Have accepted any other anti-tumor drug within 30 days before the first dose of doxorubicin hydrochloride liposome or doxorubicin;
* Pregnancy or breast feeding;
* Other situations that investigators consider as contra-indication for this study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 4 cycles (each cycle is 21 days) of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China